CLINICAL TRIAL: NCT03472833
Title: Influence of High Dose Vitamin D3 Intake on Outcome in Pancreatic Cancer Surgery: Prospective, Randomized, Open, Controlled Pilot Study
Brief Title: High-dose Vitamin D3 in Pancreas Cancer
Acronym: VITdCUT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow recruitment, patients lost to follow-up due to Covid-19 pandemic.
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VITdCUT 1.3 - 21022018
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Pancreas Cancer; Vitamin D Deficiency; Quality of Life
Keywords: V
MeSH Terms: conditions — Pancreatic Neoplasms; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose (Experimental): Intervention with high dose oral vitamin D3 supplementation.
  1 drop equals 400 I.U. This group will get 180.000 I.U. on day 1, and then 4000 I.U. per day for 60 days.
  Interventions: Drug: High-dose
- Standard-dose (Active Comparator): Intervention with standard dose oral vitamin D3 supplementation.
  1 drop equals 400 I.U. This group will get 800 I.U. per day for 60 days.
  Interventions: Drug: Standard dose

INTERVENTIONS:
Drug: High-dose — Patients will receive a high dose - 180.000 I.U. (1 drop equals 400 I.U.) of Vitamin D3 orally on day 1, and then 4000 I.U. for 60 days
  Arms: High-dose
Drug: Standard dose — Patients will receive a standard dose - 800 I.U. (equals 2 drops) of Vitamin D3 orally for 60 days
  Arms: Standard-dose

SUMMARY:
Different studies have shown that a deficiency in vitamin D (≤20ng/mL) results in higher rates in morbidity and mortality rates in cancer patients. Clinical studies investigated and demonstrated altered vitamin d tissue in pancreatic cancer. But there is no prospective study evaluating the beneficiary effects of oral supplementation of vitamin d in altered vitamin d tissue from pancreatic cancer. We want to examine the effect of a high dose vitamin D3 therapy vs. a standard base dose vitamin D3 therapy in pancreas cancer patients with a vitamin D deficiency. In case of benefit in our results we could implement vitamin D3 as a supportive standard therapy in pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

both sexes

* vitamin D deficiency(≤20ng/ml)
* patients>18 years of age
* pancreatic cancer
* surgical intervention/non-surgical intervention
* signed written informed consent

Exclusion Criteria:

* patients<18 years of age
* pregnancy
* contraindication for oral vitamin D intake
* hypercalcemia (> 2.65 mmol/l total calcium and/or > 1.35 mmol/l ionized calcium at screening)
* other ongoing vitamin D conducted trial
* known kidney stones, active tuberculosis or sarcoidosis (in the last 12 months)
* metastasized pancreatic cancer
* normal vitamin D serum levels
* missing written informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
25(OH) vitamin D | Day 60
  Blood level of Vitamin D3

SECONDARY OUTCOMES:
25(OH) vitamin D | Day 30
  Blood level of Vitamin D3
1,25(OH)2D vitamin D | Day 30
  Blood level of 1,25(OH)2D vitamin D
1,25(OH)2D vitamin D | Day 60
  Blood level of 1,25(OH)2D vitamin D
Urine Calcium | Day 30
  Calcium level in urine
Urine Calcium | Day 60
  Calcium level in urine
Osteocalcin | Day 30
  Bone marker measured in blood
Osteocalcin | Day 60
  Bone marker measured in blood
Beta-crosslaps | Day 30
  Bone marker measured in blood
Beta-crosslaps | Day 60
  Bone marker measured in blood
Calcium | Day 60
  blood measurement
Calcium | Day 30
  blood measurement
ionized calcium | Day 30
  blood measurement
ionized calcium | Day 60
  blood measurement
creatinine | Day 30
  blood measurement
creatinine | Day 60
  blood measurement
phosphate | Day 60
  blood measurement
phosphate | Day 30
  blood measurement
60-day mortality | Day 60
  Number of patients who die in the specified timeframe
hospital stay | Day 60
  Hospital stay in days
hospital readmission | Day 60
  Number of readmissions
hepcidin | Day 30
  blood level marker for iron status
hepcidin | Day 60
  blood level marker for iron status
Quality of Life questionnaire | Day 30
  evaluated by EORTC questionnaire
Quality of Life questionnaire | Day 60
  evaluated by EORTC questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kornprat, Prof. Dr., Principal Investigator — Medical University of Graz, Departement for General Surgery
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided